CLINICAL TRIAL: NCT00560261
Title: Evaluation of the Lung Capillary Blood Volume in Children With Sickle Cell Disease
Acronym: VOLCADREP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: P061013; 2007-A00913-50 (Other: ID-RCB)
Record Dates: First submitted 2007-11-16; First posted 2007-11-19 (Estimated); Last update posted 2023-02-03 (Actual); Status verified 2012-07

CONDITIONS: Sickle Cell Disease
Keywords: Sickle cell disease;; Lung capillary blood volume;; Children
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Exhalation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1:Children with sickle cell disease (Experimental): NO-CO inhalation and expiration:
  Children with sickle cell disease
  Interventions: Other: NO-CO inhalation and expiration
- 2: Healthy volunteers (Active Comparator): NO-CO inhalation and expiration:
  Healthy volunteers
  Interventions: Other: NO-CO inhalation and expiration

INTERVENTIONS:
Other: NO-CO inhalation and expiration — NO-CO inhalation and expiration
  Arms: 1:Children with sickle cell disease
Other: NO-CO inhalation and expiration — NO-CO inhalation and expiration
  Arms: 2: Healthy volunteers

SUMMARY:
Sickle cell disease (SCD) is the most common inherited disease of the world affecting African and Caribbean populations. SCD is caused by the homozygous inheritance of the gene for sickle hemoglobin (HbS). Most patients with SCD develop abnormal pulmonary function characterized by airway obstruction, restrictive lung disease, abnormal diffusing capacity, hypoxemia and pulmonary hypertension In healthy subjects, lung capillary blood volume (Qc) and membrane diffusing capacity (Dm) can be accurately measured by the nitric oxide-carbon monoxide (NO-CO) method. We propose to study, for the first time, lung capillary blood volume and alveolar membrane diffusing capacity, using the NO-CO method, in children with SCD aged of at least 6 years Early determination of lung function and pulmonary circulation in children with SCD is very important, not only for the understanding of physiopathologic mechanisms of the disease but also for a better therapeutic management of these children.

DETAILED DESCRIPTION:
We propose to study, for the first time, lung capillary blood volume and alveolar membrane diffusing capacity, using the NO-CO method, in children with SCD aged of at least 6 years. We will compare lung function and measurement of Qc and Dm in 2 groups of 120 subjects, one group of SCD children, and the other of normal children matched on age and ethnic origin. Measurement of lung capillary blood will be measured twice, to assess short term reproducibility. The measurement will be done in sitting position and lying down for one part of subjects, and at rest and during a moderate rectangular exercise for the other part of subjects. These different tests are designed to assess the physiological adaptation of pulmonary circulation in these two populations of children. Combined with complete lung function measurements, echocardiographic assessment of pulmonary hemodynamics, and measurement of exhaled nitric oxide, these evaluations will lead to a better understanding of pathophysiology of lung injury in SCD. The study will be completes at Robert Debré Hospital, in close collaboration with Sickle Cell Disease Center and Physiology Department. Children will be included after informed consent signed, as legally prescribed.

ELIGIBILITY:
Inclusion Criteria:

* Children between 6 and 18 years
* Sickle cell disease( SS,SC, SBETA O, SDpunjab) and control without sickle cell disease
* Social insurance
* Signed informed consent

Exclusion Criteria:

* Respiratory disease other tha asthma
* Cardiac disease
* Encephalopathy
* G6PD deficiency
* Consent not signed

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2008-02; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Study of lung capillary blood volume and alveolar membrane diffusing capacity using NO-CO method | The day of the measure

SECONDARY OUTCOMES:
Respiratory physiopathology's study in sickle cell disease | At the induction of the study
Valid alveolar membrane diffusing capacity using NO-CO in children with or without sickle cell disease | At the induction of the study
Purpose respiratory function follow up in sickle cell disease child | At the induction of the study
Find relationship between these vascular abnormalities and NO metabolism | At the induction of the study

CONTACTS AND LOCATIONS:
Overall Officials: Florence MISSUD, Md, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital Robert DEBRE, Paris, France

REFERENCES:
- [Result] Bokov P, Boizeau P, Pautrat J, Missud F, Ba A, Haouari Z, Denjean A, Delclaux C, Benkerrou M. Altered pulmonary capillary blood volume in childhood sickle cell disease. Eur Respir J. 2020 Dec 10;56(6):2000379. doi: 10.1183/13993003.00379-2020. Print 2020 Dec. No abstract available. PMID 32616593